CLINICAL TRIAL: NCT07254221
Title: Evaluation of Rosuvastatin Efficacy in Prevention of Anthracycline-induced Cardiac Dysfunction in Breast Cancer Patients After Chemotherapy
Brief Title: Rosuvastatin for Prevention of Anthracycline-induced Cardiac Dysfunction in Breast Cancer Patients
Acronym: ROSUBREAST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Armin Attar, Prof. Armin Attar, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IR.SUMS.MED.REC.1404.351; IRCT20191002044961N2 (Other: Iranian Registry of Clinical Trials (IRCT))
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Anthracycline-induced Cardiac Toxicity; Breast Cancer; Anthracycline Related Cardiotoxicity in Breast Cancer; Anthracycline-induced Cardiotoxicity
Keywords: Breast cancer; rosuvastatin; statin therapy,; cancer-related treatment cardiac dysfunction; anthracycline induced cardiomyopathy; cardiac dysfunction; cardiotoxicity; chemotherapy; anthracycline
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: multicenter, two-arm, double-blinded, superiority, parallel-group, randomized, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Consumption of 20 milligrams rosuvastatin daily
  Interventions: Drug: Rosuvastatin 20 mg/day
- Placebo (Placebo Comparator): Placebo (placebo tablets similar to rosuvastatin)
  Interventions: Drug: Placebo tablets similar to rosuvastatin 20mg tablets

INTERVENTIONS:
Drug: Rosuvastatin 20 mg/day — Consumption of rosuvastatin 20mg tablets every day
  Arms: Intervention
Drug: Placebo tablets similar to rosuvastatin 20mg tablets — consumption of placebo tablets similar to rosuvastatin 20mg
  Arms: Placebo

SUMMARY:
This study, called "ROSUBREAST", is a multicenter, double-blind, randomized clinical trial evaluating whether rosuvastatin (20 mg daily) can protect the heart in women with breast cancer receiving anthracycline-based chemotherapy. A total of 400 participants will be randomly assigned to receive either rosuvastatin or placebo for 12 months. The main goal is to determine whether rosuvastatin can prevent cancer treatment-related cardiac dysfunction (CTRCD), defined as a significant drop in heart pumping function. The study will also assess changes in cardiac strain, blood biomarkers, symptoms of heart failure, quality of life, and possible side effects.

DETAILED DESCRIPTION:
Introduction: Anthracycline-induced cardiotoxicity significantly threatens the long-term cardiac health of breast cancer patients undergoing chemotherapy. Statins have shown potential cardioprotective effects without compromising cancer treatment efficacy. The ROSUBREAST study aims to evaluate the efficacy of rosuvastatin in preventing CTRCD in breast cancer patients receiving anthracycline-based chemotherapy. Methods: This multicenter, two-arm, double-blinded, superiority, parallel-group, randomized, placebo controlled clinical trial will be conducted across seven oncocardiology centers in Iran. A total of 400 participants will be enrolled and will be randomly assigned in a 1:1 ratio to receive either rosuvastatin (20 mg daily) or no intervention for 12 months. The primary endpoint is the incidence of CTRCD, defined as a ≥10% reduction in left ventricular ejection fraction (LVEF) to below the lower normal limit (53%). Secondary endpoints include changes in Global Longitudinal Strain (GLS), biomarkers (Troponin, NT-proBNP, hsCRP), and development of heart failure (HF). Ancillary endpoints are quality-of-life assessments and adverse effects of treatment. Conclusion: The ROSUBREAST study seeks to provide evidence on the cardioprotective role of rosuvastatin in breast cancer patients undergoing anthracycline-based chemotherapy, potentially informing clinical guidelines and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals with ≥18 years of age
* Documented breast cancer diagnosis based on imaging and pathology findings
* Scheduled to receive the first time anthracycline-based chemotherapy

Exclusion Criteria:

* Baseline LVEF < 50%
* Prior Statin use or Statin use is indicated based on guidelines
* history of congestive heart failure (CHF) or cardiomyopathy
* Pregnancy or breastfeeding
* Unable to provide informed consent
* Unexplained persistent elevation of transaminases (>3 times upper limits of normal)
* Concomitant use of oral cyclosporine
* Metastatic invasion of cancer to other organs
* Previous cycles of chemotherapy
* Any contraindication for statin use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 400 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-04-21 (Estimated); Study Completion 2028-04-21 (Estimated)

PRIMARY OUTCOMES:
CTRCD (cancer treatment-related cardiac dysfunction) | 12 months after randomization
  CTRCD is defined as a reduction of ≥10 percentage points in LVEF by echocardiography to <53% or a >15% relative decline in global longitudinal strain (GLS) compared with baseline strain.

SECONDARY OUTCOMES:
changes in LVEF | 3, 6, and 12 months after randomization
changes in Global Longitudinal Strain (GLS) | 3, 6, and 12 months after randomization
changes in Troponin level | 3, 6, and 12 months after randomization
changes in N-terminal pro b-type Natriuretic Peptide (NT-proBNP) level | 3, 6, and 12 months after randomization
changes in High-sensitivity C-reactive Protein (hsCRP) level | 3, 6, and 12 months after randomization

OTHER OUTCOMES:
major adverse cardiovascular events (MACE) | 12 months after randomization

CONTACTS AND LOCATIONS:
Locations (7):
- Iran (7):
  - Motahari Breast Cancer Clinic, Shiraz, Fars
  - Kowsar Hospital, Fars Heart Foundation, Shiraz, Fars
  - Toba Oncology Department, Mazandaran University of Medical Sciences, Sari, Mazandaran
  - Modarres Hospital, Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province
  - Rajaee Hospital, Iran University of Medical Sciences, Tehran, Tehran Province
  - Sina Hospital, Tehran University of Medical Sciences, Tehran, Tehran Province
  - Taleghani Hospital, Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province

IPD SHARING:
Plan to Share IPD: Yes
The IPD used in the main analyses of CSR will be shared upon reasonable request from the principal investigator and confirmation by trial management committee (TMC).
Supporting Information: Study Protocol, CSR
Time Frame: The IPD can be shared after the release of CSR.
Access Criteria: Reseaonable request for IPD sharing from the principal investigator will be assessed in TMC. If the commiittee agreed and confirmed the IPD sharing, the IPD will be shared through a suitable platform.